CLINICAL TRIAL: NCT01479608
Title: A Randomized Controlled Clinical Trial to Evaluate the Benefit and Efficacy of Liver Transplantation as Treatment for Selected Patients With Liver Metastases From ColoRectal Carcinoma
Brief Title: Liver Transplantation and Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Smedman, MD, Consultant, gastrointestinal oncology, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECA-II; NCT01311453 (obsolete NCT alias)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liver Transplantation; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Transplantation or resection (randomized) (Experimental): Liver transplantation or liver resection by 1:1 randomization (open label)
  Interventions: Procedure: Liver transplantation and liver resection
- B: Liver transplantation (Experimental): For non-resectable patients metachronous disease.
  Interventions: Procedure: Liver transplantation and liver resection
- C:Liver transplantation (Experimental): For non-resectable patients synchronous disease.
  Interventions: Procedure: Liver transplantation and liver resection
- D:Liver transplantation (Experimental): For non-resectable patients synchronous disease.
  Interventions: Procedure: Liver transplantation and liver resection

INTERVENTIONS:
Procedure: Liver transplantation and liver resection

SUMMARY:
Colorectal liver metastases (CLM) are currently considered an absolute contraindication for liver transplantation (Lt) although Lt for other primary and secondary liver malignancies show excellent outcome in selected patients. Before 1995, several Lts for CLM were performed, but the outcome was poor (18% 5-year survival) and Lt for CLM was stopped. Since then, several advances have been achieved and survival following Lt has improved by almost 30%. Thus, a 5-year survival of about 50% following Lt for CLM could be anticipated.

The investigators have previously included 21 patients in a pilot study. All patients had advanced CLM at the time of Lt. Long term overall survival (OS) exceeds by far previously reported outcome for this patient group and is comparable or better than survival following repeat Lt for non-malignant diagnoses. Development of robust selection criteria may further improve the results.

The investigators will conduct a randomized controlled trial to explore whether liver transplantation in selected patients with liver metastases from CRC can obtain significant life extension and better health related quality of life compared to patients receiving surgical resection.

The investigators will also explore if patient selection according to nomo-grams for outcome of colorectal cancer can define a subgroup of patients with a 5 year survival of at least 50% or even cure from the disease.

DETAILED DESCRIPTION:
Arm D: use of extended criteria donors (ECD)

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma in colon or rectum.
* No signs of extra hepatic metastatic disease or local recurrence according to PET/CT scan.
* No signs of extra hepatic metastatic disease or local recurrence according to CT or MR (thorax/abdomen/pelvis) scan within 4 weeks prior to the faculty meeting at the transplant unit
* No signs of local recurrence judged by colonoscopy / CT colography within 12 months prior to the faculty meeting at the transplant unit
* Good performance status, ECOG 0 or 1.
* Satisfactory blood tests Hb >10g/dl, neutrophiles >1.0 (after any G-CSF), TRC >75, Bilirubin<2 x upper normal level, ASAT,ALAT<5 x upper normal level, ,Creatinine <1.25 x upper normal level. Albumin above lower normal level.
* Standard surgical procedure with adequate resection margins including circumferential resection margins (CRM) of at least ≥2mm for rectal cancer patients.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to GCP, and national/local regulations.
* Received at least 3 cycles of chemotherapy (6 weeks of treatment), with no increase in size of the lesions according to RECIST-criteria

Additional inclusion criteria for patients included in part A:

- Six or more liver metastases technically resectable

Additional inclusion criteria for patients included in part B:

* Metachronous liver metastases (more than 12 months from diagnosis of CRC and/or end of adjuvant treatment)
* Pathological classification of primary tumor as pN0 disease.
* CEA<100 ng/ml at time of primary diagnosis as well as at time of diagnosis of metastatic disease.
* Liver metastases not eligible for curative liver resection.
* Before start of 1. line chemotherapy, no lesion should be larger than 10 cm and total number of lesions should be 20 or less.
* At least 10% response (RECIST-criteria) on 1. line chemotherapy. Patients must be accepted for transplantation before progressive disease on 1. line chemotherapy.

Additional inclusion criteria for patients included in part C:

* Liver metastases not eligible for curative liver resection.
* Received 1.line treatment.
* Before start of 2. or 3. line chemotherapy, no lesion should be larger than 10 cm and total number of lesions should be 20 or less.
* At least 10% response (RECIST-criteria) on 2. or 3. line chemotherapy. Patients must be accepted for transplantation before progressive disease on 2. or 3. line chemotherapy.
* Two years or more time span from the CRC diagnosis and date of being listed on the transplantation list.

Additional inclusion criteria for patients included in part Arm D:

Patients with expected overall survival of 6-12 months without a liver transplant.

The patient might be included without further chemotherapy treatment. Patients may have resectable pulmonary lesions at time of inclusion in the present study.

Exclusion Criteria:

* Weight loss >10% the last 6 months
* Patient BMI > 30
* Other malignancies
* Prior extra hepatic metastatic disease or local relapse.
* Patients who have not received standard pre-operative, per-operative or post-operative treatment for the primary CRC.
* Palliative resection of primary CRC tumor.
* Previous randomization in this trial.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Hagness M, Foss A, Line PD, Scholz T, Jorgensen PF, Fosby B, Boberg KM, Mathisen O, Gladhaug IP, Egge TS, Solberg S, Hausken J, Dueland S. Liver transplantation for nonresectable liver metastases from colorectal cancer. Ann Surg. 2013 May;257(5):800-6. doi: 10.1097/SLA.0b013e3182823957. PMID 23360920